CLINICAL TRIAL: NCT01794260
Title: Efficacy and Safety of Topical Preparation of Essential Oil Extracted From Zingiber Cassumunar Rokb in Patients With Osteoarthritis
Brief Title: Efficacy and Safety of Topical Essential Oil Extracted From Zingiber Cassumunar Rokb in Osteoarthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFTA-01
Record Dates: First submitted 2012-12-11; First posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2012-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Moderate ot severe pain; ZINGIBER CASSUMUNAR ROXB
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo cream (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream
- Plai cream (Experimental): Cream from Zingiber cassumunar Roxb. extract
  Interventions: Drug: Cream from Zingiber cassumunar Roxb. extract

INTERVENTIONS:
Drug: Cream from Zingiber cassumunar Roxb. extract
  Arms: Plai cream
Drug: Placebo cream
  Arms: Placebo cream

SUMMARY:
The objectives of this study are to assess short term efficacy and safety of of topical preparation of essential oil extracted from ZINGIBER CASSUMUNAR ROXB in patients suffering from osteoarthritic pain

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: osteoarthritis of the knee at least on side with standard radiologic method within 6 weeks (Kellgren-Lawrence radiographic grading scale at least 1)
* Pain visual analog scale at rest at least 40 mm
* No previous analgesic treatment or receiving stable dose of analgesic drugs at least 2 weeks. If previously treated with antidepressants, glucosamine, chondroitin or diacerein, dosage should be stable for at least 3 months.
* Agree to attain non-pharmacologic treatment as prior to participate the study

Exclusion Criteria:

* having an open wound or abnormal skin at site of application
* having diagnose with other chronic arthritis such as rheumatoid arthritis
* history of allergy to the extraction of Zingiber cassumunar Roxb
* pregnancy or breastfeeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of The WOMAC (Western Ontario and McMaster Universities) index | week 8

SECONDARY OUTCOMES:
Change from baseline of Pain visual analog scale (PVAS) | week 8
Change from baseline of Global assessment of disease status (GADS) | week 8
Clinical global impression of change (CGIC) | Week 8
Patient global impression of change (PGIC) | Week 8
Adverse events | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Chuthamanee Suthisisang, Ph.D., Study Director — Department of Pharmacology, Faculty of Pharmacy, Mahidol University 447 Sri-Ayudhya Rd., Rajthevee, Bangkok 10400, Thailand; Suwimon Yeephu, M.Sc., Principal Investigator — Faculty of Pharmacy, Srinakharinwirot University; Chuthamanee Suthisisant, Ph.D, Study Chair — Mahidol University
Locations (1):
- Faculty of Medicine, Srinakharinwirot University, Ongkarak, Changwat Nakhon Nayok, Thailand